CLINICAL TRIAL: NCT04163406
Title: The Effect of Human Milk Oligosaccharides (HMOs) (2'-Fucosyllactose (2'-FL) and Lacto-N-neotetraose (LNnT)) and Galacto-oligosaccharides (GOS) on Iron Absorption From a Maize-based Porridge in Kenyan Infants
Brief Title: The Effect of Human Milk Oligosaccharides and Galacto-oligosaccharides on Iron Absorption in Kenyan Infants
Acronym: FeHMOGOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zurich (Other); Jomo Kenyatta University of Agriculture and Technology (Other); University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Principal Investigator, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FeHMOGOS
Record Dates: First submitted 2019-10-29; First posted 2019-11-14 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Anemia, Iron-deficiency
Keywords: Anemia; Iron-deficiency; Iron absorption; Prebiotic; Galacto-oligosaccharides; Human milk oligosaccharides; Infants; Kenya
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — ferrous fumarate; Health Maintenance Organizations

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ferrous fumarate (Active Comparator): Maize-based porridge fortified with iron (5mg) as ferrous fumarate
  Interventions: Dietary Supplement: ferrous fumarate
- ferrous fumarate + GOS (Active Comparator): Maize-based porridge fortified with iron (5mg) as ferrous fumarate + GOS (3g)
  Interventions: Dietary Supplement: ferrous fumarate + GOS
- ferrous fumarate + HMOs (Active Comparator): Maize-based porridge fortified with iron (5mg) as ferrous fumarate + HMOs (2'-FL (2g) + LNnT (1g))
  Interventions: Dietary Supplement: ferrous fumarate + HMOs

INTERVENTIONS:
Dietary Supplement: ferrous fumarate — Maize-based porridge fortified with iron (5mg) in form of ferrous fumarate
  Arms: ferrous fumarate
Dietary Supplement: ferrous fumarate + GOS — Maize-based porridge fortified with iron (5mg) in form of ferrous fumarate and GOS (3g)
  Arms: ferrous fumarate + GOS
Dietary Supplement: ferrous fumarate + HMOs — Maize-based porridge fortified with iron (5mg) in form of ferrous fumarate and HMOs (2'-FL (2g) + LNnT(1g))
  Arms: ferrous fumarate + HMOs

SUMMARY:
Effective and safe strategies to deliver iron to infants and young children in Sub-Saharan Africa are urgently needed. One potential strategy to improve safety of iron fortification is to limit the total amount of unabsorbed iron entering the colon by lowering the daily iron dose but at the same time ensure efficacy by maximizing absorption from this lower dose. In Kenyan infants, the investigators have recently shown that consumption of 7.5 g of the prebiotic galacto-oligosaccharides (GOS) compared to no GOS consumption increased iron absorption from an iron containing micronutrient powder by ≈60%. It is uncertain whether a lower dose of GOS can also enhance iron absorption. Another question is whether HMOs, 'natural prebiotics' found in high concentration in human breast milk, can also increase iron absorption similar to GOS. Therefore, the aim of this study is to measure fractional iron absorption from a maize-based porridge fortified with A) iron as ferrous fumarate, B) iron as ferrous fumarate and GOS and C) iron ferrous fumarate and HMOs, using an established stable iron isotope technique in 55 infants aged 8-12 months living in Msambweni and surrounding rural communities, Kwale County of southern coastal Kenya. Assessing the effect of a low dose of GOS and of HMOs on iron absorption will provide valuable information towards the development of new, highly bioavailable iron formulations for African infants.

As per the local standard of care, the participants who will be iron-deficient anemic at the end of the study will be treated with oral iron supplements. To evaluate the effects of iron supplementation on iron and anemia status and to estimate obligatory iron losses in the gastrointestinal tract, blood and fecal samples will be collected before, during and fourteen days after the beginning of the treatment with oral iron supplements. Data about the efficacy of current supplementation strategies in iron-deficient anemic children and obligatory iron losses would provide additional evidence for the optimization of iron supplementation regimens.

DETAILED DESCRIPTION:
Iron absorption from differently labelled iron-fortified maize-based test meals will be measured in 55 infants. At baseline a venipuncture blood sample will be collected from all infants for the determination of the following iron and inflammation status parameters: hemoglobin (Hb), plasma ferritin (PF), soluble transferrin receptor (sTfR), C-reactive protein (CRP) and alpha-1-acid glycoprotein (AGP), and anti-oligosaccharide immunoglobulins. Anthropometrics will be measured; demographics, the medical history and the feeding habits will be assessed using a questionnaire. A breast milk sample from all mothers will be collected for determination of HMO profile and maternal secretor status. After baseline, 30 infants will consume three different test meals on alternate days (day 1, day 3, and day 5) and 25 infants will consume two different test meals on alternate test meal days (day 1, day 3 and day 5). The order of consumption of the three test meals will be randomly assigned. Test meal A will contain 5 mg of iron as ferrous fumarate given as 2.5 mg Fe-56 and 2.5 mg Fe-54 (control test meal). Test meal B will contain 5 mg of iron as ferrous fumarate given as 2.5 mg Fe-56 and 2.5 mg Fe-58 and 4 g of GOS-75 (≈ 3 g GOS) (GOS test meal).Test meal C will contain 5 mg of iron as ferrous fumarate given as 2.5 mg Fe-56 and 2.5 mg Fe-57 and 2.0 g 2'-fucosyllactose (2'-FL) and 1.0 g lacto-N-neotetraose (LNnT) (HMO test meal). The test meals will be based on maize porridge, consisting of refined maize flour, sugar and mineral water, and will be administered between 0700 and 0900. Overnight, only breast milk will be allowed to the infant and no breast milk and no other food will be given at least 3 h before test meal administration. Test meals plus mineral water will be consumed completely in the presence of the investigators, and the infant will not be allowed to eat or drink for 2 h after the test meal. Fourteen days after the third test meal administration (day 17 and 19, respectively) a whole blood sample will be collected by venipuncture for analysis of the ratios of the different molecular weight iron incorporation into red blood cells and determination of iron and inflammation status (Hb, PF, sTfR, CRP and AGP). Furthermore, anthropometrics and some parts of the baseline questionnaire will be repeated.

At endpoint (day 17 and 19, respectively), if the infant will be diagnosed with iron-deficiency anemia (Hb concentration below 110 g/l and low red blood cells mean corpuscular volume), the caregiver will be instructed to give the infant 4mg/kg iron in the form of oral syrup, daily. Compliance during the follow-up will be assessed by weighting the iron syrup containers before and after 14 days of treatment with the iron syrup. Collection of fecal samples will be performed over 3 time periods of 72h each. The first time period will start the 3 days prior of beginning of oral iron supplementation, the second will take place on day 4, 5 and 6 of oral iron supplementation and the last on day 15, 16 and 17 of oral iron supplementation. A venepuncture blood sample will be collected in the morning after the last day of fecal sample collection (day 18 of oral iron supplementation). Furthermore, some parts of the baseline questionnaire will be repeated. Adverse events (AEs) will be assessed throughout the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Age of 8-12 months at baseline
* Assessment of good health as assessed by professional staff at Msambweni District Hospital
* The caregiver is willing to participate in the study
* The informed consent form has been read and signed by the caregiver (or has been read out to the caregiver in case of illiteracy)
* Residence in the study area for the period of the study
* Willingness of the caregiver to provide 2 blood samples from their child and 1 breast milk sample from the mother

Exclusion Criteria:

* Hb <70 g/L
* Severe wasting (Z-score weight-for-height <-3)
* Chronic or acute illness or other conditions that in the opinion of the Principle Investigator (PI) or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Participants taking part in other studies requiring the drawing of blood
* Regular intake (>2 days) of iron-containing mineral and vitamin supplements or fortified foods within the last 2 months

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption in % | Day 19
  Fractional iron absorption (%), measured as erythrocyte incorporation of stable iron isotopes at day 19

SECONDARY OUTCOMES:
Hemoglobin (Hb) | Baseline
  Iron status will be determined at baseline
Hemoglobin (Hb) | Day 19
  Iron status will be determined at day 19
Plasma Ferritin (PF) | Baseline
  Iron status will be determined at baseline
Plasma Ferritin (PF) | Day 19
  Iron status will be determined at day 19
Soluble Transferrin Receptor (sTfR) | Baseline
  Iron status will be determined at baseline
Soluble Transferrin Receptor (sTfR) | Day 19
  Iron status will be determined at day 19
C-reactive protein (CRP) | Baseline
  Inflammation status will be determined at baseline
C-reactive protein (CRP) | Day 19
  Inflammation status will be determined at day 19
Alpha-1-acid glycoprotein (AGP) | Baseline
  Inflammation status will be determined at baseline
Alpha-1-acid glycoprotein (AGP) | Day 19
  Inflammation status will be determined at day 19
Human Milk Oligosaccharides concentrations in breast milk | Baseline
  Human Milk Oligosaccharides concentrations in breast milk of the mothers of the participating infants will be measured at baseline to determine maternal secretor status.
Human Milk Oligosaccharides concentrations in breast milk | Day 19
  Human Milk Oligosaccharides concentrations in the breast milk of the mothers of the participating infants will be measured at Day 19 to determine maternal secretor status.
Anti-oligosaccharide immunoglobulins | Baseline
  Infant blood serum immunoglobulins toward mucosal oligosaccharide antigens and microbial carbohydrate antigens will be measured at baseline
Intestinal Fatty Acid Binding Protein (I-FABP) in infants diagnosed with iron deficiency anemia | Day 19
  I-FABP will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care.
Fecal calprotectin in infants diagnosed with iron deficiency anemia | 3 days before oral iron supplementation
  Fecal calprotectin will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care. Fecal calprotectin will be measured 3 days before beginning of oral iron supplementation. The sampling period will last for 72 hours.
Fecal calprotectin in infants diagnosed with iron deficiency anemia | Day 4 of oral iron supplementation
  Fecal calprotectin will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care. Fecal calprotectin will be measured on day 4 of oral iron supplementation. The sampling period will last for 72 hours.
Fecal calprotectin in infants diagnosed with iron deficiency anemia | Day 15 of oral iron supplementation
  Fecal calprotectin will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care. Fecal calprotectin will be measured on day 15 of oral iron supplementation. The sampling period will last for 72 hours.
Hemoglobin (Hb) in infants diagnosed with iron deficiency anemia | Day 18 of oral iron supplementation
  Iron status will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care
Plasma Ferritin (PF) in infants diagnosed with iron deficiency anemia | Day 18 of oral iron supplementation
  Iron status will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care
Soluble Transferrin Receptor (sTfR) in infants diagnosed with iron deficiency anemia | Day 18 of oral iron supplementation
  Iron status will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care
C-reactive protein (CRP) in infants diagnosed with iron deficiency anemia | Day 18 of oral iron supplementation
  Inflammation status will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care
Alpha-1-acid glycoprotein (AGP) in infants diagnosed with iron deficiency anemia | Day 18 of oral iron supplementation
  Inflammation status will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care
Hemoglobin in stool from infants diagnosed with iron deficiency anemia | 3 days before oral iron supplementation
  Hemoglobin concentration will be assessed in stools from infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care. Hemoglobin concentration in stools will be measured 3 days before beginning of oral iron supplementation. The sampling period will last for 72 hours.
Hemoglobin in stool from infants diagnosed with iron deficiency anemia | Day 4 of oral iron supplementation
  Hemoglobin concentration will be assessed in stools from infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care. Hemoglobin concentration in stools will be measured on day 4 of oral iron supplementation. The sampling period will last for 72 hours.
Hemoglobin in stool from infants diagnosed with iron deficiency anemia | Day 15 of oral iron supplementation.
  Hemoglobin concentration will be assessed in stools from infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care. Hemoglobin concentration in stools will be measured on day 15 of oral iron supplementation. The sampling period will last for 72 hours.
Intestinal Fatty Acid Binding Protein (I-FABP) in infants diagnosed with iron deficiency anemia | Day 18 of oral iron supplementation
  I-FABP will be assessed in infants diagnosed with iron-deficiency anaemia and receiving supplementation with oral iron syrup as per local standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof. Dr., Principal Investigator — Swiss Federal Institute of Technology
Locations (1):
- Msambweni County Referral Hospital, Msambweni, Kwale County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paganini D, Uyoga MA, Cercamondi CI, Moretti D, Mwasi E, Schwab C, Bechtler S, Mutuku FM, Galetti V, Lacroix C, Karanja S, Zimmermann MB. Consumption of galacto-oligosaccharides increases iron absorption from a micronutrient powder containing ferrous fumarate and sodium iron EDTA: a stable-isotope study in Kenyan infants. Am J Clin Nutr. 2017 Oct;106(4):1020-1031. doi: 10.3945/ajcn.116.145060. Epub 2017 Aug 16. PMID 28814396
- [Derived] Giorgetti A, Paganini D, Nyilima S, Kottler R, Frick M, Karanja S, Hennet T, Zimmermann MB. The effects of 2'-fucosyllactose and lacto-N-neotetraose, galacto-oligosaccharides, and maternal human milk oligosaccharide profile on iron absorption in Kenyan infants. Am J Clin Nutr. 2023 Jan;117(1):64-72. doi: 10.1016/j.ajcnut.2022.10.005. Epub 2022 Dec 15. PMID 36789945